CLINICAL TRIAL: NCT00738582
Title: An Open-Label Clinical Trial of MORAb-009 in Combination With Pemetrexed and Cisplatin in Subjects With Mesothelioma
Brief Title: An Efficacy Study of MORAb-009 (Amatuximab) in Subjects With Pleural Mesothelioma
Acronym: Amatuximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-009-003 Amatuximab; 2008-005448-18 (EudraCT Number); NCT00923455 (obsolete NCT alias)
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2015-11

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — amatuximab; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Pemetrexed, Cisplatin and MORAb-009 (Amatuximab)
  Interventions: Drug: MORAb-009 (Amatuximab); Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: MORAb-009 (Amatuximab) — MORAb-009 (Amatuximab) by IV on Days 1 and 8 every 21 days for 6 cycles.
Drug: Pemetrexed — Pemetrexed 500 mg/m2 on Day 1 of each 21-day cycle for 6 cycles
Drug: Cisplatin — Cisplatin 75 mg/m2 on Day 1 of each 21-day cycle for 6 cycles

SUMMARY:
This research is being done to find out if pemetrexed and cisplatin work better when given together with an experimental drug called MORAb-009 in patients with malignant pleural mesothelioma.

ELIGIBILITY:
Primary Inclusion Criteria:

* Confirmed diagnosis of malignant pleural mesothelioma (MPM) with the following characteristics: unresectable disease (or otherwise not a candidate for curative surgery); epithelial type or biphasic (mixed) type with low sarcomatous content.
* Measurable disease at Screening by computed tomography (CT)(or magnetic resonance imaging [MRI]).
* KPS of greater than or equal to 70% at Screening.
* Life expectancy of at least 3 months

Primary Exclusion Criteria:

* Sarcomatous type of mesothelioma
* Prior systemic therapy or radiotherapy for MPM; local radiotherapy for symptom control (ie, non-curative intent) is permitted.
* Confirmed presence of CNS tumor involvement.
* Evidence of other active malignancy requiring treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-12-31 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2014-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wallin, MD, Study Director — Morphotek
Locations (28):
- United States (12):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Diego, La Jolla, California
  - UCLA Medical Hematology & Oncology, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Christiana Care Health System, Newark, Delaware
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University--Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - NIH/National Cancer Institute, Bethesda, Maryland
  - Columbia University Medical Center, New York, New York
  - Mary Babb Randolph Cancer Center, Morgantown, West Virginia
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Laval, Quebec, PQ
- Germany (7):
  - HELIOS Klinikum Emil von Behring, Berlin
  - Asklepios Fachkliniken Müchen-Gauting, Gauting
  - Krankenhaus Großhansdorf, Großhansdorf
  - Asklepios Klinik Harburg, Hamburg
  - Medizinsche Hochschule Hannover, Hanover
  - Fachklinik für Lungenerkrankungen Immenhausen, Immenhausen
  - Medizinische Klinik (Hämatologie/Onkologie), München
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede
  - Erasmus MC, Rotterdam
- Spain (5):
  - H. de la Santa Creu i Sant Pau, Barcelona
  - Consorci Sanitari Parc Taulí, Barcelona
  - H. Son Dureta, Palma de Mallorca
  - Clínica Universitaria de Navarra, Pamplona
  - H. Virgen del Rocío, Seville

RESULTS

PARTICIPANT FLOW:
Groups:
- Amatuximab/Pemetrexed/Cisplatin: Participants received amatuximab 5 milligram per kilogram (mg/kg), Intravenous (IV) infusion on Days 1 and 8 with pemetrexed 500 milligram per meter square (mg/m^2), IV infusion on Day 1 and cisplatin 75 mg/m^2, IV infusion on Day 1 of each 21-day cycle for approximately 6 cycles during combination therapy (Cycle length is 21 days).
- Amatuximab: Participants who completed 6 cycles of combination therapy or who discontinued chemotherapy because of intolerable toxicity continued receiving single agent amatuximab 5 mg/kg, IV infusion on Day 1 and 8 of each 21-day cycle until disease progression or death for all subsequent cycles (up to 52 Cycles) (Cycle length is 21 days).
Period: Combination Therapy
Arm/Group | Amatuximab/Pemetrexed/Cisplatin | Amatuximab
Started | 89 | 0
Completed | 56 | 0
Not Completed | 33 | 0
Not completed — Completed Combination Therapy | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Toxicity to Chemotherapy | 1 | 0
Not completed — Other | 5 | 0
Not completed — Adverse Event | 16 | 0
Not completed — Progressive Disease | 9 | 0
Period: Maintenance Therapy
Arm/Group | Amatuximab/Pemetrexed/Cisplatin | Amatuximab
Started | 0 (This arm ended once all participants entered into the Maintenance Therapy phase of the study.) | 56 (Only eligible participants entered into this phase of the study.)
Completed | 0 | 0
Not Completed | 0 | 56
Not completed — Other | 0 | 2
Not completed — Adverse Event | 0 | 6
Not completed — Progressive Disease | 0 | 47
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants received amatuximab 5 mg/kg, IV infusion on Days 1 and 8 with pemetrexed 500 mg/m^2, IV infusion on Day 1 and cisplatin 75 mg/ m^2, IV infusion on Day 1 of each 21-day cycle for approximately 6 cycles during combination therapy. Participants who completed 6 cycles of combination therapy or who discontinued chemotherapy because of intolerable toxicity continued receiving single agent amatuximab 5 mg/kg, IV infusion on Day 1 and 8 of each 21-day cycle until disease progression or death for all subsequent cycles (up to 52 Cycles [Cycle length is 21 days]).
Arm/Group | All Participants
Number analyzed (Participants) | 89
Age, Continuous [Median (Full Range); unit: Years] | 67 [46 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival (PFS) Responders and Non-responders at Month 6
Description: Number of participants with PFS responders and non-responders at Month 6 was reported. PFS was defined as the time from the date of the first dose of amatuximab to the date of disease progression or death due to any cause, as determined by independent radiologist based on the modified Response Evaluation Criteria in Solid Tumors (RECIST) utilizing the total tumor measurement (performed by computerized tomography (CT)/magnetic resonance imaging (MRI)) which includes the pleural unidimensional measure plus the total of the target lesion(s) measurement. A "response", in terms of PFS, was defined to be at least a 6-month stabilization of disease. Progressive disease (PD) as measured by Modified RECIST was defined as an increase of at least 20 percent (%) in the total tumor measurement over the nadir measurement, or the appearance of one or more new lesions.
Time Frame: Month 6
Population: Primary Efficacy Population: all participants who received at least 1 dose of amatuximab and met key eligibility criteria (had measurable disease at screening, had unresectable disease, and had at least 1 response assessment or died after starting treatment with amatuximab). Here, number of participants analyzed are first 77 enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 77
Participants
  PFS Responders | 26
  PFS non-responders | 51

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR, defined as the percentage of participants with objective evidence of complete response (CR) or partial response (PR) as determined by independent radiologist based on the modified RECIST utilizing the total tumor measurement (performed by CT/ MRI) which includes the pleural unidimensional measure plus the total of the target lesion(s) measurement. Tumor assessments performed up to the initiation of further anticancer therapy were considered. CR was defined as the disappearance of all target lesions with no evidence of tumor elsewhere, and PR was defined as at least a 30% reduction in the total tumor measurement. A confirmed response required a repeat observation on two occasions 4 weeks apart. ORR = CR + PR.
Time Frame: From the date of first dose until evidence of CR or PR, up to approximately 5 years
Population: Primary Efficacy Population: all participants who received at least 1 dose of amatuximab and met key eligibility criteria (had measurable disease at screening, had unresectable disease, and had at least 1 response assessment or died after starting treatment with amatuximab).
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 84
Percentage of participants | 34.5

3. Secondary Outcome: Duration of Response (DR)
Description: DR was derived for those participants who achieved a PFS Response and had an objective evidence of CR or PR. DR was defined as the time (in months) from first documentation of objective response (CR or PR) to the first documentation of disease progression or death [as determined by independent radiologist based on the modified RECIST utilizing the total tumor measurement (performed by CT/ MRI) which includes the pleural unidimensional measure plus the total of the target lesion(s) measurement]. Tumor assessments performed up to the initiation of further anticancer therapy were considered. CR was defined as the disappearance of all target lesions with no evidence of tumor elsewhere, and PR was defined as at least a 30% reduction in the total tumor measurement. PD as measured by Modified RECIST was defined as an increase of at least 20% in the total tumor measurement over the nadir measurement, or the appearance of one or more new lesions.
Time Frame: From the first documentation of objective response (CR or PR) to the first documentation of disease progression, up to approximately 5 years
Population: Primary Efficacy Population: all participants who received at least 1 dose of amatuximab, met key eligibility criteria (had measurable disease at screening, had unresectable disease, and had at least 1 response assessment or died after starting treatment with amatuximab). Here, number of participants analysed included responders (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 29
Months | 9.2 [6.0 to 16.2]

4. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR was derived for those participants with objective evidence of CR or PR. TTR was defined as the time from the date of the first dose of amatuximab to first documentation of objective tumor response. CR was defined as the disappearance of all target lesions with no evidence of tumor elsewhere, and PR was defined as at least a 30% reduction in the total tumor measurement.
Time Frame: From the date of the first dose to first documentation of objective response, up to approximately 5 years
Population: Primary Efficacy Population: all participants who received at least 1 dose of amatuximab and met key eligibility criteria (had measurable disease at screening, had unresectable disease, and had at least 1 response assessment or died after starting treatment with amatuximab). Here, number of participants analysed included responders (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 29
Months | 2.3 [2.1 to 3.8]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of amatuximab to the date of death.
Time Frame: From the date of first dose to the date of death, up to approximately 5 years
Population: Safety population consisted of all participants who received at least 1 dose of amatuximab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 89
Months | 14.8 [12.4 to 18.8]

6. Secondary Outcome: Overall Progression Free Survival
Description: Overall PFS was defined as the time from the date of first dose of amatuximab to the date of disease progression or death due to any cause. In the absence of confirmation of death, the survival time was censored at the date of the last follow-up contact. Tumor assessments performed up to the initiation of further anticancer therapy were considered. PD as measured by Modified RECIST was defined as an increase of at least 20% in the total tumor measurement over the nadir measurement, or the appearance of one or more new lesions.
Time Frame: From the date of first dose of amatuximab to the date of disease progression, up to approximately 5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 84
Months | 6.3 [6.0 to 7.8]

7. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Amatuximab
Description: An adverse event (AE) was any untoward medical occurrence (example; any unfavorable and unintended sign including abnormal laboratory findings, symptom or disease) in a participant or clinical investigation participant after providing written informed consent for participation in the study until the end of study visit. TEAEs were defined as an AE that developed or worsened in severity during the on-treatment period (from first dose of amatuximab to 30 days after last dose of amatuximab). SAE was defined as any adverse event (appearance of [or worsening of any pre-existing]) undesirable sign, symptom or medical conditions which is fatal or life-threatening or results in persistent or significant disability/incapacity or constitutes a congenital anomaly/birth defect or requires inpatient hospitalization or prolongation of existing hospitalization or is medically significant.
Time Frame: From date of first dose of study drug up to 30 days after the last dose of study treatment, up to approximately 5 years
Population: Safety population included all participants who received at least 1 dose of amatuximab.
Measure: Count of Participants; unit: Participants
Groups:
- Amatuximab/Pemetrexed/Cisplatin: Participants received amatuximab 5 mg/kg, IV infusion on Days 1 and 8 with pemetrexed 500 mg/m^2, IV infusion on Day 1 and cisplatin 75 mg/ m^2, IV infusion on Day 1 of each 21-day cycle for approximately 6 cycles during combination therapy (Cycle length is 21 days).
- Amatuximab: Participants who completed 6 cycles of combination therapy or who discontinued chemotherapy because of intolerable toxicity continued receiving single agent amatuximab 5 mg/kg, IV infusion on Day 1 and 8 of each 21-day cycle until disease progression or death for all subsequent cycles (up to 52 Cycles [Cycle length is 21 days]).
Arm/Group | Amatuximab/Pemetrexed/Cisplatin | Amatuximab
Number analyzed (Participants) | 89 | 56
Participants
  Participants with at least 1 TEAE | 89 | 52
  Participants with at least 1 SAE | 38 | 15

ADVERSE EVENTS:
Time Frame: From date of first dose of study drug up to 30 days after the last dose of study treatment, up to approximately 5 years
Arm/Group | Amatuximab/Pemetrexed/Cisplatin | Amatuximab
All-Cause Mortality (participants affected / at risk) | 4/89 | 0/56
Serious Adverse Events (participants affected / at risk) | 38/89 | 15/56
Other Adverse Events (participants affected / at risk) | 89/89 | 52/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amatuximab/Pemetrexed/Cisplatin (N=89) | Amatuximab (N=56)
Vertigo (Ear and labyrinth disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Infectious peritonitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pyopneumothorax (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 2 | 1
Non-cardiac Chest Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Infusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Atrial Fibrillation (Cardiac disorders) | 4 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Cardio-respiratory Arrest (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Cystitis Radiation (Injury, poisoning and procedural complications) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Hypersensitivity (Immune system disorders) | 4 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Peripheral Embolism (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
C-reactive Protein Increased (Investigations) | 1 | 0
International Normalised Ratio Increased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient Ischemic Attack (Nervous system disorders) | 0 | 1
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amatuximab/Pemetrexed/Cisplatin (N=89) | Amatuximab (N=56)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 1
Abdominal Tenderness (Gastrointestinal disorders) | 1 | 1
Anal Fissure (Gastrointestinal disorders) | 1 | 0
Anorectal Discomfort (Gastrointestinal disorders) | 1 | 0
Bowel Movement Irregularity (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 2
Salivary Hypersecretion (Gastrointestinal disorders) | 1 | 0
Tongue Coated (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Oesophageal Pain (Gastrointestinal disorders) | 0 | 1
Oedema Mouth (Gastrointestinal disorders) | 0 | 1
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 63 | 14
Constipation (Gastrointestinal disorders) | 28 | 4
Vomiting (Gastrointestinal disorders) | 28 | 9
Diarrhoea (Gastrointestinal disorders) | 25 | 4
Stomatitis (Gastrointestinal disorders) | 12 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 11 | 5
Dyspepsia (Gastrointestinal disorders) | 9 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 7 | 1
Flatulence (Gastrointestinal disorders) | 5 | 0
Abdominal Distension (Gastrointestinal disorders) | 4 | 2
Abdominal Pain (Gastrointestinal disorders) | 4 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 0
Dry Mouth (Gastrointestinal disorders) | 2 | 0
Eructation (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 52 | 11
Asthenia (General disorders) | 16 | 6
Non-Cardiac Chest Pain (General disorders) | 16 | 13
Oedema Peripheral (General disorders) | 15 | 7
Chills (General disorders) | 13 | 5
Pyrexia (General disorders) | 13 | 3
Mucosal Inflammation (General disorders) | 6 | 0
Catheter Site Pain (General disorders) | 3 | 0
Chest Discomfort (General disorders) | 3 | 2
Chest Pain (General disorders) | 3 | 0
Pain (General disorders) | 3 | 1
General Physical Health Deterioration (General disorders) | 2 | 0
Oedema (General disorders) | 2 | 1
Catheter Site Swelling (General disorders) | 1 | 0
Extravasation (General disorders) | 1 | 0
Face Oedema (General disorders) | 1 | 0
Feeling Hot (General disorders) | 1 | 0
Feeling Jittery (General disorders) | 1 | 0
Injection Site Reaction (General disorders) | 1 | 0
Medical Device Complication (General disorders) | 1 | 1
Pre-Existing Condition Improved (General disorders) | 1 | 0
Catheter Site Haemorrhage (General disorders) | 0 | 1
General Symptoms (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 40 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 2
Hyponatremia (Metabolism and nutrition disorders) | 8 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 17 | 3
Dizziness (Nervous system disorders) | 15 | 3
Headache (Nervous system disorders) | 11 | 5
Paraesthesia (Nervous system disorders) | 6 | 5
Neuropathy Peripheral (Nervous system disorders) | 4 | 10
Polyneuropathy (Nervous system disorders) | 3 | 3
Hypoaesthesia (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 2 | 0
Ageusia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Balance Disorder (Nervous system disorders) | 1 | 0
Dysaethesia (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Parosmia (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1
Phrenic Nerve Paralysis (Nervous system disorders) | 1 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 1 | 0
Restless Legs Syndrome (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 1 | 1
Sinus Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Vascular Headache (Nervous system disorders) | 1 | 0
Burning Sensation (Nervous system disorders) | 0 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 1
Dizziness Postural (Nervous system disorders) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 26 | 3
Neutropenia (Blood and lymphatic system disorders) | 26 | 2
Leukopenia (Blood and lymphatic system disorders) | 10 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 14 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 5 | 2
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Scar Pain (Skin and subcutaneous tissue disorders) | 2 | 1
Skin Discolouration (Skin and subcutaneous tissue disorders) | 2 | 2
Cold Sweat (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Penile Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Facial Wasting (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 7
Candidiasis (Infections and infestations) | 4 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 4
Cellulitis (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 3 | 2
Respiratory Tract Infection (Infections and infestations) | 3 | 1
Rhinitis (Infections and infestations) | 3 | 1
Bronchitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1
Device Related Infection (Infections and infestations) | 1 | 0
Eye Infection (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 1
Herpes Virus Infection (Infections and infestations) | 1 | 0
Herpes Zoster Opthalmic (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Oral Candidiasis (Infections and infestations) | 1 | 0
Oral Herpes (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia Primary Atypical (Infections and infestations) | 1 | 0
Pyopneumothorax (Infections and infestations) | 1 | 0
Tinea Pedis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3
Influenza (Infections and infestations) | 0 | 2
Appendictis (Infections and infestations) | 0 | 1
Febrile Infection (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Infectious Peritonitis (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 1
Weight Decreased (Investigations) | 17 | 3
Blood Creatinine Increased (Investigations) | 14 | 2
Breathe Sounds Abnormal (Investigations) | 6 | 0
Haemoglobin Decreased (Investigations) | 6 | 1
White Blood Cell Count Decreased (Investigations) | 5 | 1
Platelet Count Decreased (Investigations) | 4 | 0
Weight Increased (Investigations) | 4 | 0
Blood Urea Increased (Investigations) | 3 | 0
C-Reactive Protein Increased (Investigations) | 2 | 1
Neutrophil Count Decreased (Investigations) | 2 | 0
Percussion Test Abnormal (Investigations) | 2 | 0
Blood Albumin Decreased (Investigations) | 1 | 0
Blood Cholesterol Increased (Investigations) | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0
Blood Phosphorus Decreased (Investigations) | 1 | 0
Blood Potassium Decreased (Investigations) | 1 | 0
Blood Sodium Decreased (Investigations) | 1 | 0
Cardiac Murmur (Investigations) | 1 | 0
Glomerular Filteration Rate Decreased (Investigations) | 1 | 0
Heart Rate Irregular (Investigations) | 1 | 0
International Normalised Ratio Increased (Investigations) | 1 | 1
Occult Blood Positive (Investigations) | 1 | 0
White Blood Cell Count Increased (Investigations) | 1 | 0
Anion Gap Increased (Investigations) | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1
Blood Bicarbonate Increased (Investigations) | 0 | 1
Blood Lactate Dehyrogenase Increased (Investigations) | 0 | 1
Gamma Glutamyl Transferase Increased (Investigations) | 0 | 1
Red Blood Cell Count Decreased (Investigations) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 5
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 4 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Plantar Fascitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Lacrimation Increased (Eye disorders) | 9 | 1
Vision Blurred (Eye disorders) | 4 | 1
Conjunctivitis (Eye disorders) | 3 | 1
Dry Eye (Eye disorders) | 2 | 1
Diplopia (Eye disorders) | 1 | 0
Erythema Of Eyelid (Eye disorders) | 1 | 0
Eye Irritation (Eye disorders) | 1 | 1
Eye Pruritus (Eye disorders) | 1 | 0
Eye Swelling (Eye disorders) | 1 | 0
Eyelid Oedema (Eye disorders) | 1 | 0
Lacrimal Disorder (Eye disorders) | 1 | 0
Periorbital Oedema (Eye disorders) | 1 | 0
Scleral Haemorrhage (Eye disorders) | 1 | 0
Visual Impairement (Eye disorders) | 1 | 0
Vitreous Floaters (Eye disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 11 | 2
Vertigo (Ear and labyrinth disorders) | 7 | 1
Deafness (Ear and labyrinth disorders) | 1 | 2
Deafness Bilateral (Ear and labyrinth disorders) | 1 | 0
Dysacusis (Ear and labyrinth disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Ototoxicity (Ear and labyrinth disorders) | 1 | 1
Hypertension (Vascular disorders) | 6 | 5
Hypotension (Vascular disorders) | 5 | 0
Flushing (Vascular disorders) | 2 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Hot Flush (Vascular disorders) | 1 | 1
Pallor (Vascular disorders) | 1 | 0
Peripheral Coldness (Vascular disorders) | 1 | 0
Peripheral Embolism (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Varicose Vein (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Embolism Venous (Vascular disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 7 | 2
Depression (Psychiatric disorders) | 3 | 0
Restlessness (Psychiatric disorders) | 3 | 0
Sleep Disorder (Psychiatric disorders) | 3 | 1
Depressed Mood (Psychiatric disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 0
Bulimia Nervosa (Psychiatric disorders) | 1 | 0
Confusion State (Psychiatric disorders) | 1 | 0
Panic Attack (Psychiatric disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 6 | 2
Atrial Fibrillation (Cardiac disorders) | 5 | 2
Palpitations (Cardiac disorders) | 4 | 1
Bradycardia (Cardiac disorders) | 2 | 1
Tachyarrhythmia (Cardiac disorders) | 2 | 0
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 7 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 0
Eye Injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 2
Limb Injury (Injury, poisoning and procedural complications) | 0 | 2
Cystitis Radiation (Injury, poisoning and procedural complications) | 0 | 1
Radiation Oesophagitis (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Hypersensitivity (Immune system disorders) | 11 | 2
Drug Hypersensitivity (Immune system disorders) | 3 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Glycosuria (Renal and urinary disorders) | 1 | 0
Ketonuria (Renal and urinary disorders) | 1 | 0
Micturition Urgency (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Renal Pain (Renal and urinary disorders) | 1 | 0
Renal Tubular Necrosis (Renal and urinary disorders) | 1 | 1
Urine Flow Decreased (Renal and urinary disorders) | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Pelvic-Ureteric Obstruction (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Neoplasm of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Neoplasm of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balanitis (Reproductive system and breast disorders) | 1 | 0
Breast Pain (Reproductive system and breast disorders) | 1 | 0
Epidifymitis (Reproductive system and breast disorders) | 1 | 0
Genital Burning Sensation (Reproductive system and breast disorders) | 1 | 0
Genital Pain (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Breast Swelling (Reproductive system and breast disorders) | 0 | 1
Colectomy (Surgical and medical procedures) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other